CLINICAL TRIAL: NCT02633969
Title: A Phase IIA, Open-label, Safety and Pharmacokinetic Study of Indomethacin Capsules in Pediatric Subjects 6 to <17 Years of Age With Mild to Moderate Acute Postoperative Pain Following Elective Surgery
Brief Title: Study of Indomethacin Capsules to Treat Pain Following Surgery in Children Ages 6 to <17 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Iroko Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IND2-15-08
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Indomethacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indomethacin Capsules low dose (Experimental): Indomethacin Capsules low dose twice daily for up to three days
  Interventions: Drug: Indomethacin Capsules low dose
- Indomethacin Capsules high dose (Experimental): Indomethacin Capsules high dose twice daily for up to three days
  Interventions: Drug: Indomethacin Capsules high dose

INTERVENTIONS:
Drug: Indomethacin Capsules low dose
  Arms: Indomethacin Capsules low dose
Drug: Indomethacin Capsules high dose
  Arms: Indomethacin Capsules high dose

SUMMARY:
The purposes of this study are to evaluate the safety and tolerability and to model the single-dose pharmacokinetic profile of indomethacin capsules low dose and high dose in children ages 6 to <17 years experiencing mild to moderate acute postoperative pain.

DETAILED DESCRIPTION:
This was a phase IIA, multicenter, open-label, fixed-dose study. The study consisted of 3 periods: a Screening Period (Day -14 to Day -1, Preoperative Visit), a Treatment Period (Days 1-3), and a Follow-Up Period (Days 4-14).

Informed consent from the subject's legally authorized representative (parent/guardian) and assent (as applicable) from the subject were obtained before the subject underwent any protocol-specified procedures or assessments. Screening/Baseline data (including medical history, vital signs, physical examination, and clinical laboratory tests) were collected for each subject and used for initial assessment of eligibility. Clinical laboratory test results obtained before screening were acceptable for determining eligibility if they were collected within 1 week before the Screening/Baseline Visit. Subjects must have met all study entry criteria to be eligible for enrollment. To adequately assess the safety and tolerability of administering multiple doses of Tivorbex Capsules in this population, subjects who were likely to require multiple-day treatment for pain (preferably for the full 3-day treatment period) were enrolled.

As part of screening, subjects were required to demonstrate the ability to swallow a placebo capsule that corresponded in size to the study drug dose for their body weight. Eligible subjects were required to refrain from taking prohibited medications throughout the study. Prohibited analgesic medications taken at the time of the Screening/Baseline Visit were discontinued 12 hours before the first dose of study drug (perioperative analgesic/anesthetic medications given during the surgical procedure were exempt from this restriction) and were captured in the appropriate electronic case report form (eCRF).

Rescue medication as part of the postoperative treatment regimen was permitted according to the local standard of care unless contraindicated for use with Tivorbex. Subjects could receive the first dose of Tivorbex any time after surgery, following discontinuation of intravenous (IV) analgesics, oral opioids, or acetaminophen.

Subjects received the first dose of study drug at the site on Day 1. Four blood samples for PK analysis were collected at various time points via indwelling catheter over the first 12 hours after initial dosing.

After the last blood sample collection (ie, up to approximately 12 hours after dosing), if treatment for mild to moderate pain was still needed, the second dose of study drug was administered. Subjects were instructed to continue dosing as needed up to twice daily for up to 3 days (through Day 3) or until treatment for pain was no longer needed, whichever came first.

Subjects remained at the study site until the last blood sample for drug concentration measurement was obtained in the 8- to 12-hour time interval after the first dose of study drug and were discharged at the discretion of the investigator. Depending on the nature of the pediatric surgical procedure, subjects could be managed as inpatients (possibly for the entire duration of the study) or as outpatients according to the standard of care required to treat the subject's condition. Upon discharge from the site, the parent/guardian was given a diary and instructed to record dates/times of study drug administration and concomitant medications (including rescue medication use). Inpatients did not require a diary because this information was captured in hospital or site records. Before discharge from the site, a supply of study drug was dispensed to the subject's parent/guardian.

On Day 1 of the Treatment Period (Day 1 to Day 3), the investigator reviewed Screening/Baseline Visit assessments (including adverse events [AEs] and concomitant medications, vital signs, physical examination, and entry criteria) and clinical laboratory test results. Following surgery, subjects who continued to meet study entry criteria had their pain severity assessed. Pain severity for children ages 6 to <12 years was assessed using the FPS R. Pain severity for children ages ≥12 years was assessed using a 0 to 10 NRS. All subjects were to have a baseline FPS-R score or baseline NRS of >0 and <7 to be eligible for the study.

Subjects contributed 4 blood samples for PK analysis from 1 of the 2 sampling schemes as follows:

Sampling Scheme #1 Sampling Scheme #2 0.15 to 0.75 hours 0.75 to 1.25 hours 1.25 to 2.25 hours 1.75 to 3.0 hours 3.0 to 6.0 hours 6.0 to 8.0 hours 8.0 to 10.0 hours 10.0 to 12.0 hours

If a subject experienced inadequate pain relief or increasing pain or severe pain following Tivorbex treatment, the investigator could consider administration of additional postoperative analgesic treatment (ie, "rescue medication") according to applicable standards of care. During study participation, the subject was to refrain from taking any other NSAIDs, aspirin, or opioid combination products containing NSAIDs or aspirin. If the pain experienced by a subject continued to be unacceptable following rescue medication administration, the investigator was to consider withdrawing the subject from the study.

Subjects returned to the site for a Final Visit approximately 7 days (± 3 days) after the final dose of Tivorbex. During this visit, a physical examination was performed, vital signs were assessed, and subject diaries were collected and reviewed. The study drug was accounted for and unused study drug was collected. All AE data were reviewed and recorded. Any ongoing AE was followed to a satisfactory resolution, until the subject became stable, or until the event could be explained by another known cause(s) (ie, concurrent condition or medication) and clinical judgment indicated that further evaluation was not warranted.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥20 kilograms
* Mild to moderate acute pain requiring treatment with analgesic medication
* Willing to have blood samples taken for PK sampling using an indwelling catheter
* Must be able to swallow capsules and can tolerate oral medication
* For females: is not of reproductive potential (defined as premenarchal) or is practicing an acceptable method of birth control

Exclusion Criteria:

* Severe acute pain
* Chronic analgesic or glucocorticoid use for any condition within 6 months before dosing with study drug
* Emergency surgery
* History of allergic reaction, hypersensitivity, or clinically significant intolerance to indomethacin, aspirin, codeine, acetaminophen, or any NSAID
* History of peptic ulcer disease or a GI event (eg, perforation, obstruction, or bleed) within 6 months before screening
* Current use of any medication that may cause a clinically significant drug interaction when co-administered with indomethacin
* Current use of any medication that might affect the pharmacokinetics of indomethacin
* History of bleeding disorders
* Developmental delay or behavioral problems that would make it difficult to assess pain
* Impaired liver function
* Clinically significant renal or cardiovascular disease
* Any medical condition that compromises ability to swallow, absorb, metabolize, or excrete the study drug
* Previously received any investigational product or device within 30 days before Screening or scheduled to receive an investigational device or another investigational drug (other than that in this study) during the course of this study
* Previous participation in this clinical study or currently taking indomethacin

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Plasma Concentrations of indomethacin | 0-12 hours after first dose of indomethacin
  The estimated typical value for clearance (tvCL) following a single indomethacin dose based on population pharmacokinetic (PopPK) modeling using sparse plasma concentration data in pediatric subjects.

SECONDARY OUTCOMES:
Safety of Indomethacin Capsules low dose and high dose as assessed by the incidence of adverse events from baseline to Day 3 or early termination | Baseline to Day 3/Early Termination
  Tivorbex Capsules 20 mg and 40 mg were generally well tolerated. No deaths or SAEs were reported. Overall, 6 subjects (20.0%) experienced at least 1 TEAE during the study. All TEAEs were mild in intensity and 2 TEAEs (1 in each treatment group) of vomiting were considered to be related to the study drug.
  The most common TEAEs were vomiting (13.3%) and nausea (6.7%). Vomiting and nausea were the only TEAEs reported in >1 subject in either group. The frequency of nausea and vomiting observed in this study is consistent with the findings from previous pediatric studies on NSAIDs.No gastrointestinal AEs commonly reported with NSAIDs, such as bleeding, ulceration, or perforation of the stomach and intestines were reported, nor were cardiovascular thrombotic events.No AEs of acute-type allergic reaction or bronchospasm were reported.
  Vital sign and physical examination findings did not reveal any safety concerns; specifically no new onset hypertension was observed during the study.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Sheffield, Alabama
  - Aurora, Colorado
  - Coral Gables, Florida
  - Durham, North Carolina
  - Orem, Utah